CLINICAL TRIAL: NCT05068115
Title: An Study on the Trend of Change and Influencing Factors of Clinicopathologic Characteristics, Diagnosis and Treatment Pattern, and Survival Status of Young Breast Cancer in China
Brief Title: Characteristics and Treatment Trends of Young Breast Cancer in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Peng Yuan, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: NCC2985
Record Dates: First submitted 2021-08-15; First posted 2021-10-05 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Therapeutics; Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Young breast cancer patients in China from 2000 to 2015, of whom the clinical features, diagnosis and treatment models and survival status are described.
  Interventions: Procedure: Clinical characteristics, diagnosis and treatment, survival status

INTERVENTIONS:
Procedure: Clinical characteristics, diagnosis and treatment, survival status — Describe the clinical characteristics, diagnosis and treatment, survival status and the trends of young breast cancer
  Other Names: This is a retrospective study to observe and describe the diagnosis and treatment of previous young breast cancer patients without intervention

SUMMARY:
To describe the clinical characteristics, the diagnosis and treatment, the survival status and change trend of young breast cancer patients in China from 2000 to 2015, and to explore and discuss the main influencing factors.

DETAILED DESCRIPTION:
In this study, medical records and follow-up information of young breast cancer patients (age ≤35 years at first diagnosis) who were first diagnosed and treated in the years (2000, 2003, 2006, 2009, 2012 and 2015) were collected from multiple hospitals in China from 2000 to 2015, to establish a retrospective cohort of young breast cancer patients. Clinical characteristics, diagnosis and treatment, and survival rates of young breast cancer patients from 2000 to 2015 were analyzed. To explore the main factors affecting the clinical diagnosis and treatment and the survival of patients.

ELIGIBILITY:
Inclusion Criteria:

* Young Breast cancer patients (≤35 years old) in China

Exclusion Criteria:

* Breast cancer patients (>35 years old) in China

Ages: 18 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: Young Breast cancer patients (≤35 years old) in China
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Clinical features and trend | Between 2000 and 2015
  To describe the clinical characteristics and trends of young breast cancer patients in China
Diagnosis and treatment and trend | Between 2000 and 2015
  To describe the methods of diagnosis and treatment in young breast cancer patients in China and the changing trend, to explore the main factors affecting diagnosis and treatment
Survival situation and change trend | Between 2000 and 2015
  To describe the survival and change trend of young breast cancer patients in China, to explore the main factors affecting the prognosis of young breast cancer patients